CLINICAL TRIAL: NCT02088190
Title: Effect of Aging on Bariatric Surgery-induced Changes in Metabolism and Cognition
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO-235
Record Dates: First submitted 2014-03-11; First posted 2014-03-14 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Insulin Resistance; Cognitive Impairment
MeSH Terms: conditions — Insulin Resistance; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Age group 1: Age > 60 years old
  Interventions: Procedure: Sleeve gastrectomy
- Age group 2: Age < 60 years old
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Type of bariatric surgery

SUMMARY:
The investigators hypothesize that the improvements in insulin sensitivity, beta (β)-cell function, and inflammation will be greater, and the improvement in sarcopenic obesity will be less, in younger versus older individuals after substantial weight loss induced by sleeve gastrectomy bariatric surgery.

DETAILED DESCRIPTION:
With an aging population that is increasingly susceptible to obesity and obesity-related comorbidities including sarcopenia and diabetes, effective and safe treatment options tailored to the needs of older adults are imperative. While medication and lifestyle interventions generally fail to achieve sustained large-scale weight loss, bariatric surgery is the most effective long-term weight loss treatment for obese patients and improves many of the medical complications associated with obesity. Sleeve gastrectomy (SG) results in substantial weight loss and may be more appropriate for older adults due to its low rate of complications and mortality. Therefore, SG has been proposed as a reasonable primary treatment modality in older obese individuals, with a substantial recent increase in the number of interventions performed. Despite the potential benefits, very little is known of the physiologic and metabolic effects of bariatric surgery, including SG, on glucose homeostasis and muscle physiology in older adults. A fundamental understanding of the effects of excess adiposity and weight loss interventions is of profound importance, especially with emerging evidence that earlier treatment of obesity may delay/prevent many comorbidities. An underlying inflammatory state has been implicated in the pathogenesis of sarcopenia and insulin resistance and may provide an important connection to the age-related declines seen in older obese patients. Therefore, this study aims to evaluate the modifying effect of age and inflammation on the SG-induced changes in body composition, muscle physiology, and insulin sensitivity. This protocol will be conducted in two age cohorts (greater than 60 and less than 50 years old).

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 yrs old
* BMI ≥ 35 kg/m2
* Undergoing laparoscopic sleeve gastrectomy (SG)

Exclusion Criteria:

* Smokers
* Presence of diabetes mellitus
* Taking any medication that might affect metabolism
* Severe organ dysfunction
* Pregnant or breastfeeding
* Prior gastrointestinal surgery that might affect study results
* Unable or unwilling to follow the study protocol or any reason the research team believes the subject is not an appropriate candidate for this study
* Weight >450 pounds (Will be unable to fit on the DXA scanner)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo laparoscopic sleeve gastrectomy (SG) at The Ohio State University (OSU) Wexner Medical Center will be divided into two cohorts: 1). Greater than or equal to 60 years of age and 2). Less than 60 years of age.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2018-11 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity | Change from baseline in Insulin sensitivity at 15% weight loss (up to 4 months after surgery)
  Subjects will undergo a clamp procedure to assess insulin sensitivity at baseline and 15% weight loss after surgery

SECONDARY OUTCOMES:
Change in Beta cell function | Change from baseline to 15% weight loss (up to 4 months after surgery)
  Subjects will undergo a mixed meal tolerance test at baseline and 15% weight loss

CONTACTS AND LOCATIONS:
Overall Officials: David P Bradley, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No